CLINICAL TRIAL: NCT01003418
Title: Safety and Immunogenicity Study of GSK Biologicals' Pandemic Influenza Candidate Vaccine (GSK2340272A) in Children Aged 8 to 12 Weeks
Brief Title: Study to Evaluate Safety and Immunogenicity of GSK Biologicals' Pandemic Influenza (H1N1) Candidate Vaccine in Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prematurely for logistic reasons, not related to safety or efficacy of the vaccine.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113629
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-09

CONDITIONS: Influenza
Keywords: GSK2340272A; H1N1 pandemic influenza
MeSH Terms: conditions — Influenza, Human | interventions — Heptavalent Pneumococcal Conjugate Vaccine

ARMS (2):
- GSK2340272A Group 1 (Experimental): Healthy male or female children, between and including 8 and 12 weeks of age at the time of first vaccination, received 2 primary doses of GSK2340272A vaccine, according to a 0-28 day schedule. Subjects also received routine infant immunisation (Infanrix™-IPV/Hib) and Prevenar™ vaccine at Day 14, Month 3 and Month 10. All vaccines were administered intramuscularly into the anterolateral region of the thigh.
  Interventions: Biological: GSK2340272A GSK Biologicals' investigational influenza pandemic vaccine; Biological: Infanrix™-IPV/Hib; Biological: Prevenar
- GSK2340272A Group 2 (Experimental): Healthy male or female children, between and including 8 and 12 weeks of age at the time of first vaccination, received 2 primary doses of GSK2340272A vaccine, according to a 0-4 month schedule. Subjects also received routine infant immunisation (Infanrix™-IPV/Hib) and Prevenar™ vaccine at Day 14, Month 3 and Month 10. All vaccines were administered intramuscularly into the anterolateral region of the thigh.
  Interventions: Biological: GSK2340272A GSK Biologicals' investigational influenza pandemic vaccine; Biological: Infanrix™-IPV/Hib; Biological: Prevenar

INTERVENTIONS:
Biological: GSK2340272A GSK Biologicals' investigational influenza pandemic vaccine — Two doses; intramuscular administration
Biological: Infanrix™-IPV/Hib — Routine infant immunisation vaccine, three doses administered intramuscularly
Biological: Prevenar — Routine infant immunisation vaccine, three doses administered intramuscularly

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of two doses of the H1N1 candidate vaccine administered in children aged between 8 and 12 weeks at the time of first vaccination.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LARs) can and will comply with the requirements of the protocol
* Children, male or female, aged between 8 and 12 weeks at the time of first study vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Healthy children, as established by medical history and clinical examination when entering the study.
* Parent/LAR with access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device.
* Born after a gestation period of >= 36 to <= 42 weeks.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If ANY exclusion criterion applies, the subject must not be included in the study:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Acute disease at the time of enrolment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing required).
* History of any neurological disorders or seizures.
* A family history of congenital or hereditary immunodeficiency.
* Receipt of systemic glucocorticoids within one month of study enrolment, or any other cytotoxic or immunosuppressive drug since birth.
* Administration of any vaccines within two weeks before study enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study.
* Previous administration of any H1N1 vaccine, of any seasonal influenza vaccine.
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis, Haemophilus influenzae type b, and/or Streptococcus pneumoniae with the exception of vaccines where the first dose can be given within the first two weeks of life according to the national recommendations.
* History of intercurrent diphtheria, tetanus, pertussis, poliomyelitis, Haemophilus influenzae type b disease.
* Major congenital defects or serious chronic illness.
* Child in care.
* Any known or suspected allergy to any constituent of the influenza, DTPa-IPV/Hib and pneumococcal study vaccines; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza, DTPa-IPV/Hib and pneumococcal vaccine.

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2009-11-17 (Actual); Primary Completion 2010-11-25 (Actual); Study Completion 2010-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Norway (4):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Hønefoss
  - GSK Investigational Site, Lierskogen
  - GSK Investigational Site, Oslo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113629 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 8 subjects were enrolled in the study as the study was terminated prematurely for logistic reasons, not related to safety or efficacy of the vaccine.
Pre-assignment Details: Subjects who were enrolled completed the study but the lack of data due to the small enrollment number prevented any statistical analyses to be performed. No statistical analyses were performed as per planned in the protocol. All study results summarized below are based solely on individual data listings generated.
Groups:
- GSK2340272A Group 1: Healthy male or female children, between and including 8 and 12 weeks of age at the time of first vaccination, received 2 primary doses of GSK2340272A vaccine, according to a 0-28 day schedule. Subjects also received routine infant immunisation (Infanrix-IPV/Hib) and Prevenar vaccine at Day 14, Month 3 and Month 10. All vaccines were administered intramuscularly into the anterolateral region of the thigh.
- GSK2340272A Group 2: Healthy male or female children, between and including 8 and 12 weeks of age at the time of first vaccination, received 2 primary doses of GSK2340272A vaccine, according to a 0-4 month schedule. Subjects also received routine infant immunisation (Infanrix-IPV/Hib) and Prevenar vaccine at Day 14, Month 3 and Month 10. All vaccines were administered intramuscularly into the anterolateral region of the thigh.
Period: Overall Study
Arm/Group | GSK2340272A Group 1 | GSK2340272A Group 2
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340272A Group 1 | GSK2340272A Group 2 | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Full Range); unit: Weeks] | 9 [7 to 10] | 8 [7 to 9] | 8.63 [7 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Arabic/North African heritage | 1 | 0 | 1
  White-Caucasian/European heritage | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Solicited Local or General Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Assessed solicited general symptoms were drowsiness, fever, irritability and loss of appetite.
Time Frame: During the 7-days post-Dose 1 period (Days 0-6)
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group 1 | GSK2340272A Group 2
Number analyzed (Participants) | 5 | 3
Participants
  Pain | 2 | 0
  Redness | 2 | 0
  Swelling | 2 | 0
  Drowsiness | 3 | 1
  Fever | 1 | 0
  Irritability | 3 | 1
  Loss of appetite | 0 | 1

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities/crying that cannot be comforted. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 2-weeks post-Dose 1 period (Days 0-13)
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group 1 | GSK2340272A Group 2
Number analyzed (Participants) | 5 | 3
Participants
  Any AE(s) | 2 | 2
  Grade 3 AE(s) | 0 | 0
  Related AE(s) | 0 | 0

3. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed included medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: During the 2-weeks post-Dose 1 period (Days 0-13)
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group 1 | GSK2340272A Group 2
Number analyzed (Participants) | 5 | 3
Participants | 0 | 0

4. Secondary Outcome: Number of Subjects With Any Solicited Local or General Symptoms
Description: as for outcome 1
Time Frame: During the 7-days post-Dose 2 period (Days 28 + 7 days for Group 1; Month 4 + 7 days for Group 2)
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group 1 | GSK2340272A Group 2
Number analyzed (Participants) | 5 | 3
Participants
  Pain | 3 | 0
  Redness | 1 | 1
  Swelling | 2 | 3
  Drowsiness | 5 | 3
  Fever | 3 | 2
  Irritability | 3 | 2
  Loss of appetite | 2 | 1

5. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited AEs
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any AE reported in addition to those solicited during the clinical study. Also any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited AE. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities/crying that cannot be comforted. Related = AE assessed by the investigator as related to the vaccination. Results about unsolicited AEs for this endpoint were based on individual listings.
Time Frame: During the 28-day (Days 0-27) follow-up period after each study vaccine administration
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group 1 | GSK2340272A Group 2
Number analyzed (Participants) | 5 | 3
Participants
  Any AE(s) | 3 | 2
  Grade 3 AE(s) | 0 | 0
  Related AE(s) | 0 | 0

6. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed included medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. Results about SAEs were based on individual listings.
Time Frame: During the entire study period (From Month 0 up to Month 11)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group 1 | GSK2340272A Group 2
Number analyzed (Participants) | 5 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: within the 7-day (Days 0-6) follow-up period after each study vaccination. Unsolicited AEs: within the 28-day (Days 0-27) follow-up period after each study vaccination. SAEs: throughout the entire study period (from Month 0 up to Month 11).
Arm/Group | GSK2340272A Group 1 | GSK2340272A Group 2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2340272A Group 1 (N=5) | GSK2340272A Group 2 (N=3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tracheal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Pain (General disorders) | 4 | 0
Redness (General disorders) | 2 | 1
Swelling (General disorders) | 2 | 3
Drowsiness (General disorders) | 5 | 3
Fever (General disorders) | 4 | 2
Irritability (General disorders) | 4 | 3
Loss of appetite (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.